CLINICAL TRIAL: NCT06899815
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effects of Single and Multiple Administration of F230 Tablets in Healthy Adult Volunteers
Brief Title: Preliminary Human Trials of F230 Tablets
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDN-F230-202401
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAD single dose group (Experimental): A total of 6 dose groups A1-A6: F230 are initially expected to be developed (A1-A6 test groups were administered 3mg, 6mg, 12mg, 20mg, 30mg, 40mg, respectively). The specific incremental dose can be adjusted according to the test situation. The A1 dose group included 8 volunteers (stratified by sex, F230 tablets: placebo =3:1), and the A2 to A6 dose group included 14 volunteers (stratified by sex, F230 tablets: Placebo =6:1), F230 tablets or placebo were taken orally on an empty stomach on the day of administration. From the night before the start of the trial to the end of the trial evaluation period (A1:D-1 ~ D3/A2-A6:D-1 ~ D2), the volunteers were kept in the phase I research room. During the study period, safety assessment and PK biological sample collection were conducted according to the protocol. The volunteers completed a safety check on day 3(A1)or day2(A2-A6).
  Interventions: Drug: F230 tablets
- MAD multiple dose group (Experimental): It is preliminarily expected to carry out 3 dose groups, preset 6mg, 12mg, 20mg, the frequency of administration will be determined according to the results of a single administration test, continuous administration for 7 days. 14 volunteers were included in each group (stratified by sex, F230 tablets: placebo = 6:1), and a total of 42 volunteers were planned to be included. All volunteers were in the research center from the day before administration (D-1) to 24h after the last administration (D8). During the study period, safety assessment and PK biological sample collection were conducted according to the protocol. On the 8th day of the study (D8, 24h after the last administration), the procedures prescribed in the protocol and related safety checks were completed, and they could leave the research center after comprehensive evaluation by the researchers. The volunteers then returned to the study center on day 9 (D9,48h after the last dose) or for safety follow-up.
  Interventions: Drug: F230 tablets
- Research on the effects of food on drugs (Experimental): It is planned to include 16 volunteers. A stratified block randomization method was adopted, with gender as the stratification factor. Volunteers were randomly assigned to two drug administration sequence groups (K-C group and C-K group), with 8 cases in each group. That is, 8 volunteers were administered on an empty stomach in the first cycle, and the other 8 volunteers were administered within half an hour after consuming a high-fat meal in the first cycle and eluted on the second day (D2). After a total of 3 days (72 hours) of elution, the volunteers received the second cycle of administration on the 6th day (D6). Volunteers who received the drug on an empty stomach in the first cycle were given the drug within half an hour after a high-fat meal. Volunteers who received the drug after a high-fat meal in the first cycle were given the drug on an empty stomach. Complete the procedures stipulated in the plan and related safety checks on the 7th day of the study.
  Interventions: Drug: F230 tablets

INTERVENTIONS:
Drug: F230 tablets — SAD： A1: F230 tablets 3mg;A2: F230 tablets 6mg;A3: F230 tablets 12mg;A4: F230 tablets 20mg;A5: F230 tablets 30mg;A6: F230 tablets 40mg .
  MAD： B1: F230 tablets 6mg; B2: F230 tablets 12mg; B3: F230 tablets 20mg; Studies on the effects of food on drugs:Group K-C: The first cycle was fasting administration, and the second cycle was postprandial administration;C-K:The first cycle was given after meals, and the second cycle was given on an empty stomach.

SUMMARY:
F230 is a new Class 1 chemical drug jointly developed by Beijing Contini Pharmaceutical Co., Ltd. for the treatment of pulmonary hypertension (Notification number: 2024LP01242, 2024LP01243). The in vitro activity and in vivo toxicology tests of F230, the lead compound for the treatment of PAH developed by Beijing Contini Pharmaceutical Co., LTD., showed that F230 had the same in vitro activity as the endothelin antagonist on the market. The pharmacodynamics of F230 in rats with nephrogenic hypertension induced by Sunitinib showed that F230 could reduce proteinuria and improve renal index.It is expected to bring higher treatment and survival benefits to the corresponding patients. According to the spirit of NMPA new drug approval, on the basis of the completion of preclinical studies of this drug, the safety, tolerability and pharmacokinetic characteristics of single administration and multiple administration of this drug in healthy volunteers should be investigated first, and the influence of food on the pharmacokinetic characteristics of F230 in humans should be investigated, so as to recommend a safe and effective administration regimen for phase II clinical trials.

DETAILED DESCRIPTION:
This study consists of three parts: the first part is a single administration study (SAD test), the second part is a multiple administration study (MAD test), and the third part is a Food Effect study, which is divided into multiple cohorts according to dose groups and administration regimens.

Single Administration Trial (SAD) : This randomized, double-blind, placebo-controlled, dose-increasing, single-center clinical study was designed to evaluate the safety, tolerability, and pharmacokinetic profile of F230 single administration in healthy volunteers. A total of 78 healthy adult volunteers were planned to be included.This part is expected to develop 6 dose groups: 3mg, 6mg, 12mg, 20mg, 30mg, 40mg, and the groups are indicated by A1-A6. Group A1 planned to include 8 healthy volunteers (stratified by sex, A1:F230 tablets: placebo =3:1), and group A2-A6 planned to include 14 healthy volunteers (stratified by sex, F230 tablets: placebo =6:1), increasing from the initial dose group to the maximum dose group, with each group receiving only a single dose.Qualified volunteers who met the inclusion criteria and did not meet the exclusion criteria were admitted to the phase I laboratory one day before the experiment (D-1) and randomly grouped. The researchers conducted education on the environment, regulations, etc., unified dinner, fasting after 21:00, and did not refrain from drinking water. On the day of administration, F230 tablets or placebo were taken orally on an empty stomach. From the night before the start of the trial to the end of the trial evaluation period (A1:D-1 ~ D3/A2-A6:D-1 ~ D2), the volunteers were kept in the phase I research room. During the study period, safety assessment and PK biological sample collection were conducted according to the protocol. Volunteers completed a safety check on day 3(A1)/ day 2(A2-A2-A6), and were allowed to leave the study center after a comprehensive assessment by the investigator, and then returned to the study center onday 4(A1)/ day 3(A2-A2-A6) or by telephone for safety follow-up.

Multiple dose trial (MAD) : This randomized, double-blind, placebo-controlled, dose-increasing, single-center clinical study was designed to evaluate the safety, tolerability, and pharmacokinetics of multiple dose F230 tablets in healthy volunteers. 42 healthy adult volunteers were scheduled to participate.

According to the preliminary results of the SAD study, this study is expected to carry out 3 dose groups: 6 mg, 12mg and 20mg groups are represented by B1, B2 and B3, and the administration frequency is determined according to the SAD test results for 7 consecutive days. 14 volunteers are included in each dose group (stratified by sex, F230 tablets: placebo =6:1).Qualified volunteers who met both the inclusion criteria and did not meet any of the exclusion criteria were admitted to the Phase I research room 1 day before the experiment (D-1) and randomly grouped. The researchers conducted education on the environment, regulations, etc., unified dinner, and fasting after 21:00 without drinking water. The volunteers were given F230 tablets or placebo orally on an empty stomach in the morning, and the frequency of administration was determined according to the SAD test results, and they were given continuously for 7 days. All volunteers were in the research center from the day before administration (D-1) to 48h after the last administration (D8). During the study period, safety assessment and PK biological sample collection were conducted according to the protocol, and the procedures prescribed in the protocol and related safety checks were completed on the 9th day of the study (D8, 24h after the last administration). The volunteers were allowed to leave the study center after a comprehensive assessment by the investigator, and then returned to the study center on day 9 (D9, 48h after the last dose) or by telephone for safety follow-up.

Research on the Effect of Food on Drugs:

This part is a randomized, open, two-cycle, double-cross clinical study design, referred to as the food impact study. According to the preliminary results of SAD study, it is expected to carry out a dose group: X mg, and a total of 16 healthy volunteers are planned to be included. The volunteers are randomly divided into K-C and C-K groups by stratified block randomization method, taking gender as a stratified factor, and are randomly divided into two groups at 1:1 ratio, with 8 cases in each group.

Qualified volunteers who met both the inclusion criteria and did not meet any of the exclusion criteria were admitted to the Phase I research room 1 day before the experiment (D-1) and randomly grouped. The researchers conducted education on the environment, regulations, etc., unified dinner, and fasting after 21:00 without drinking water. In the first cycle, K-C group was given fasting, C-K group was given within half an hour after eating a high-fat meal, and group exit examination was conducted on day 2 (D2). After 3 days (72h) of elution, the volunteers underwent a second cycle of dosing on day 6 (D6). In the second cycle, K-C group was administered within half an hour after eating a high-fat meal, and C-K group was administered on an empty stomach. Safety assessment and PK biological sample collection will be conducted during the study in accordance with protocol requirements.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following criteria to be selected:

1. Healthy volunteers, half male and half female, should be replaced by volunteers of the same sex;
2. Age: 18 ~ 45 years old;
3. Weight: male ≥50kg, female ≥45kg, 19≤BMI≤26 (BMI= weight (kg)/height 2 (m2));
4. Pass the comprehensive health examination: vital signs, physical examination, blood urine routine, blood pregnancy, blood glucose, blood lipid, blood electrolyte, hepatitis B surface antigen, liver and kidney function, hepatitis C, HIV and syphilis antibody test, 12-lead electrocardiogram, nicotine, urine drug screening, alcohol breath test, abdominal B-ultrasound, chest X-ray examination, etc., no abnormalities or abnormalities have no clinical significance;
5. Before participating in the study, have a detailed understanding of the nature, significance, possible benefits, possible inconveniences and potential dangers of the trial, and voluntarily participate in this clinical trial, can communicate well with the investigators, comply with the requirements of the entire study, and have the ability to understand and sign the written informed consent.

Exclusion Criteria:

* Volunteers who meet one of the following conditions are not eligible for this study:

  1. Participants in any other clinical trial within three months prior to the trial;
  2. Serum ALT > upper limit of normal (ULN), AST > Upper limit of normal (ULN), TBil > upper limit of normal (ULN);
  3. (Consultation) whether there are underlying liver diseases, such as chronic hepatitis B, chronic hepatitis C, alcoholic liver disease and non-alcoholic fatty liver disease, and cirrhosis;
  4. (Consultation) Have any disease that may affect the safety of the trial or the process of the drug in vivo, including but not limited to: Heart, liver, kidney, endocrine, digestive, immune, respiratory, nervous or psychiatric systems, or other pre-existing or existing diseases of the above systems [especially cardiovascular disease including those at risk for cardiovascular disease, any gastrointestinal disease that interferes with drug absorption (e.g. symptoms of irritable bowel syndrome, history of inflammatory bowel disease), active pathological bleeding (e.g. peptic ulcer), urticaria, epilepsy, epilepsy, etc. Sensitive rhinitis, eczematous dermatitis, asthma, active pulmonary tuberculosis, etc.
  5. (Consultation) Allergy: If there is a history of drug, food allergy or skin allergy;
  6. (Interview) Any drug that inhibits or induces liver metabolism of the drug in the 28 days prior to the use of the study drug (common liver enzyme inducers: barbiturates such as phenobarbital, carbamazepine, aminomide, grofulvin, methylaminopropyl, phenytoin, Grumette, rifampin, dexamethasone; Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide);

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Single dose:PK parameters: Cmax | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: Tmax | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: AUC0-t | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: AUC0-∞ | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: t1/2 | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: λz | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: Vz/F | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: CL/F | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: AUC_%Extrap | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: MRT | Within 48 hours of dosing
  Blood PK parameters
Single dose:PK parameters: Ae_u (t1-t2) | Within 48 hours of dosing
  Urine PK parameters
Single dose:PK parameters: Ae_u (0-t) | Within 48 hours of dosing
  Urine PK parameters
Single dose:PK parameters: Rate_u (max) | Within 48 hours of dosing
  Urine PK parameters
Single dose:PK parameters:Fe_u (0-t) | Within 48 hours of dosing
  Urine PK parameters
Multiple administration: PK parameters:Cmax,ss | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters:Tmax,ss | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: AUC0-τ,ss | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: AUC0-t | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: AUC0-∞ | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters:Cmin,ss | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: Cav,ss | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: t1/2 | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: λz | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: CLss/F | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: AUC_%Extrap | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: MRT | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: DF | Within 48 hours of dosing
  Blood PK parameters
Multiple administration: PK parameters: Rac | Within 48 hours of dosing
  Blood PK parameters
Effects of food on single pharmacokinetic parameters: Cmax | Within 48 hours of dosing
  Blood PK parameters
Effects of food on single pharmacokinetic parameters: Tmax | Within 48 hours of dosing
  Blood PK parameters
Effects of food on single pharmacokinetic parameters: AUC | Within 48 hours of dosing
  Blood PK parameters

SECONDARY OUTCOMES:
Safety and tolerance assessment:Adverse event | SAD: 3 days
  Adverse events (AE) are all adverse medical events that occur after a clinical study volunteer receives an investigational drug. It may present as symptoms, signs, disease, or abnormalities in laboratory tests, but may not have a causal relationship with the investigational drug. An AE can be an aggravation of an existing disease, symptoms, signs, laboratory abnormalities, or a newly diagnosed disease, newly occurring symptoms, signs, laboratory outliers, etc.
Safety and tolerance assessment:Adverse event | MAD: 9 days
  Adverse events (AE) are all adverse medical events that occur after a clinical study volunteer receives an investigational drug. It may present as symptoms, signs, disease, or abnormalities in laboratory tests, but may not have a causal relationship with the investigational drug. An AE can be an aggravation of an existing disease, symptoms, signs, laboratory abnormalities, or a newly diagnosed disease, newly occurring symptoms, signs, laboratory outliers, etc.
Safety and tolerance assessment:Adverse event | Effects of food on drugs test: 9 days
  Adverse events (AE) are all adverse medical events that occur after a clinical study volunteer receives an investigational drug. It may present as symptoms, signs, disease, or abnormalities in laboratory tests, but may not have a causal relationship with the investigational drug. An AE can be an aggravation of an existing disease, symptoms, signs, laboratory abnormalities, or a newly diagnosed disease, newly occurring symptoms, signs, laboratory outliers, etc.
Safety and tolerance assessment:Vital signs measurement：temperature | SAD: 3 days;
  Measure the axillary temperature, the normal value is 35.9-36.7℃
Safety and tolerance assessment:Vital signs measurement：temperature | MAD: 9 days
  Measure the axillary temperature, the normal value is 35.9-36.7℃
Safety and tolerance assessment:Vital signs measurement：temperature | Effects of food on drugs test: 9 days
  Measure the axillary temperature, the normal value is 35.9-36.7℃
Safety and tolerance assessment:Vital signs measurement：breathing | SAD: 3 days
  Adult resting breathing rate 12-20 beats per minute
Safety and tolerance assessment:Vital signs measurement：breathing | MAD: 9 days
  Adult resting breathing rate 12-20 beats per minute
Safety and tolerance assessment:Vital signs measurement:breathing | Effects of food on drugs test: 9 days
  Adult resting breathing rate 12-20 beats per minute
Safety and tolerance assessment:Vital signs measurement:blood pressure | SAD: 3 days
  Systolic and diastolic blood pressure were measured
Safety and tolerance assessment:Vital signs measurement:blood pressure | MAD: 9 days
  Systolic and diastolic blood pressure were measured
Safety and tolerance assessment:Vital signs measurement:blood pressure | Effects of food on drugs test: 9 days
  Systolic and diastolic blood pressure were measured
Safety and tolerance assessment:12-lead ECG test/holter ECG | SAD: 3 days
  A 12-lead ECG is a non-invasive test that records the heart's electrical activity through 12 electrodes placed on the body surface. Includes 6 limb leads (Ⅰ, Ⅱ, Ⅲ, aVR, aVL, aVF) and 6 chest leads (V1-V6).A Holter ECG uses a portable device to continuously record heart activity over 24-48 hours, capturing transient abnormalities during daily activities or symptom episodes.It includes PR interval, QRS wave group, QT interval, ST segment,and PP/RR interval.
Safety and tolerance assessment:12-lead ECG test/holter ECG | MAD: 9 days
  A 12-lead ECG is a non-invasive test that records the heart's electrical activity through 12 electrodes placed on the body surface. Includes 6 limb leads (Ⅰ, Ⅱ, Ⅲ, aVR, aVL, aVF) and 6 chest leads (V1-V6).A Holter ECG uses a portable device to continuously record heart activity over 24-48 hours, capturing transient abnormalities during daily activities or symptom episodes.It includes PR interval, QRS wave group, QT interval, ST segment,and PP/RR interval
Safety and tolerance assessment:12-lead ECG test/holter ECG | Effects of food on drugs test: 9 days
  A 12-lead ECG is a non-invasive test that records the heart's electrical activity through 12 electrodes placed on the body surface. Includes 6 limb leads (Ⅰ, Ⅱ, Ⅲ, aVR, aVL, aVF) and 6 chest leads (V1-V6).A Holter ECG uses a portable device to continuously record heart activity over 24-48 hours, capturing transient abnormalities during daily activities or symptom episodes.It includes PR interval, QRS wave group, QT interval, ST segment,and PP/RR interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Hubei, Wuhan, China

IPD SHARING:
Plan to Share IPD: No